CLINICAL TRIAL: NCT01263223
Title: Effect of LY2216684 on Ambulatory Heart Rate and Blood Pressure in Patients With Major Depressive Disorder Who Are Being Treated With Selective Serotonin Reuptake Inhibitors
Brief Title: A Study of LY2216684 in Major Depressive Disorder in Patients Taking Selective Serotonin Reuptake Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12607; H9P-EW-LNCP (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684, placebo, LY or placebo (Experimental): Period 1: 18 milligrams (mg) LY2216684 administered orally once daily on Days 1-4
  Period 2: placebo administered orally once daily on Days 1-4
  Period 3: 36 mg LY2216684 or placebo administered orally daily on Days 1-4
  Interventions: Drug: LY2216684; Drug: Placebo
- Placebo, LY2216684, placebo or LY (Experimental): Period 1: placebo administered orally once daily on Days 1-4
  Period 2: 18 mg LY2216684 administered orally once daily on Days 1-4
  Period 3: 36 mg LY2216684 or placebo administered orally daily on Days 1-4
  Interventions: Drug: LY2216684; Drug: Placebo

INTERVENTIONS:
Drug: LY2216684 — Administered orally
Drug: Placebo — Administered orally

SUMMARY:
The purpose of this study is to determine the effect of LY2216684 on heart rate and blood pressure in research participants with MDD who are being treated with an SSRI (selective serotonin reuptake inhibitors). Information about any side effects that may occur will also be collected. The duration of participation in this study is approximately 24 days not including the screening visit. This study requires 1 clinic confinement of 17 days/16 nights and 1 Follow-up Outpatient Visit. A screening visit is required within 30 days prior to the start of the study. In both periods 1 and 2, the study involves 4 single daily doses of 18 mg LY2216684 or placebo taken as 2 tablets by mouth. In period 3, the study involves four single daily doses of 36 mg LY2216684 or placebo taken as 4 tablets by mouth.

ELIGIBILITY:
Inclusion Criteria:

* Are patients that have been diagnosed with major depressive disorder (MDD) and are on a stable dose of an selective serotonin reuptake inhibitor (SSRI) for at least 4 weeks prior to enrollment, as determined by medical history and physical examination.
* Male patients: Agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug.
* Female patients: Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or Women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause for at least 1 year without menses or 6 months without menses and a follicle stimulating hormone (FSH) >40 milli-international-units/milliliter (mIU/mL).
* Have a body mass index (BMI) of up to 32.0 kilogram/squaremeter (kg/m2).
* Have normal blood pressure (BP) and pulse rate (systolic BP <140, diastolic BP <90; supine position and standing) as determined by the investigator.
* Patients that have a diagnosis of hypertension but are well controlled on a stable dose (at least 4 weeks of diuretic, angiotensin converting enzyme [ACE]-inhibitor, or angiotensin 2 receptor inhibitor) are acceptable for inclusion in this study. Allowance of a specific anti-hypertensive is per the investigator's discretion.
* Have screening clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to any compound related to LY2216684.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684.
* Have a clinically significant abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a significant history of or presence of cardiovascular (including dysrhythmias), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders, or any condition capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have unequal BP (> 20 millimeter of mercury [mm Hg]) in the left arm versus right arm (as measured with a BP cuff) or have absent or unequal radial pulses in either arm.
* Have a history of seizure disorders.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Use of over-the-counter or prescription medication (other than stable doses of SSRI as noted above) with a narrow therapeutic index (including, but not limited to warfarin or clopidogrel) or those that are known to have an effect on heart rate (e.g., beta-blockers) within 14 days prior to dosing.
* Use of any drugs or substances that are known to be a strong inducer or inhibitor of cytochrome P450 2D6 (CYP2D6) or cytochrome P450 3A4 (CYP3A4) within 30 days prior to check-in (study entry) and during the conduct of the study.
* Have donated blood of more than 500 milliliter (mL) within 4 weeks prior to screening.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to check-in (study entry)until the completion of the study (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any patients unwilling to adhere to study caffeine restrictions.
* Patients must adhere to the smoking restrictions of the Clinical Research Unit (CRU) while a resident of the CRU.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment or are unwilling to avoid during the study.
* Have a documented or suspected history of glaucoma.
* Patients determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 18-mg LY2216684; Placebo; 36-mg LY2216684 or Placebo: Period 1: 18-milligram (mg) LY2216684 (LY) administered orally once daily on Days 1-4
  Period 2: Placebo administered orally, once daily on Days 1-4
  Period 3: 36-mg LY2216684 or Placebo administered orally, once daily on Days 1-4
- Placebo; 18-mg LY2216684; Placebo or 36-mg LY2216684: Period 1: Placebo administered orally, once daily on Days 1-4
  Period 2: 18-mg LY2216684 administered orally, once daily on Days 1-4
  Period 3: 36-mg LY2216684 or Placebo administered orally, once daily on Days 1-4
Period: Period 1
Arm/Group | 18-mg LY2216684; Placebo; 36-mg LY2216684 or Placebo | Placebo; 18-mg LY2216684; Placebo or 36-mg LY2216684
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: 3-Day Washout
Arm/Group | 18-mg LY2216684; Placebo; 36-mg LY2216684 or Placebo | Placebo; 18-mg LY2216684; Placebo or 36-mg LY2216684
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | 18-mg LY2216684; Placebo; 36-mg LY2216684 or Placebo | Placebo; 18-mg LY2216684; Placebo or 36-mg LY2216684
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 3
Arm/Group | 18-mg LY2216684; Placebo; 36-mg LY2216684 or Placebo | Placebo; 18-mg LY2216684; Placebo or 36-mg LY2216684
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: 7-day Follow-up
Arm/Group | 18-mg LY2216684; Placebo; 36-mg LY2216684 or Placebo | Placebo; 18-mg LY2216684; Placebo or 36-mg LY2216684
Started | 12 | 11
Completed | 11 (One participant who did not complete received Placebo in Period 3.) | 10 (One participant who did not complete received 36-mg LY2216684 in Period 3.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Overall Study Participants: Period 1: 18-mg LY2216684 or Placebo administered orally, once daily on Days 1-4.
  Period 2: Participants who received LY2216684 in Period 1, then received Placebo administered orally, once daily on Days 1-4 in Period 2. Participants who received Placebo in Period 1, then received 18-mg LY2216684 administered orally, once daily on Days 1-4 in Period 2.
  Period 3: 36-mg LY2216684 or Placebo administered orally, once daily on Days 1-4.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum and Mean Change From Baseline in Ambulatory Heart Rate on Day 1
Description: Heart rate was determined during ambulatory blood pressure monitoring (ABPM). Mean pre-dose ABPM values from Day 1 in Period 1 were used as baseline. Maximum and mean changes in ABPM heart rate were determined from a 24-hour continuous ABPM monitoring for Day 1 (0 to 24 hours). Least Squares (LS) mean changes from baseline were calculated with a mixed effects model including sequence, period, study day, treatment groups, and interaction between treatment groups and study day as fixed effects, and subject as random effect.
Time Frame: Baseline through the 24-hour interval on Day 1
Population: All participants with a baseline observation and at least 1 post-baseline observation on Day 1 were included in the analyses. Observations with 18-mg LY2216684 included Periods 1 and 2. Observations with Placebo included Periods 1, 2, and 3. Therefore, some participants contributed 2 Placebo observations to the overall data.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Units Other Than Participants: Observations
Groups:
- 18-mg LY2216684: Participants received a single, oral dose of 18-mg LY2216684 each day over 4 days.
- Placebo: Participants received a single, oral dose of Placebo each day over 4 days.
Arm/Group | 18-mg LY2216684 | Placebo
Number analyzed (Participants) | 23 | 23
Number analyzed (Observations) | 23 | 27
beats per minute (bpm)
  Mean Change | 13.3 [9.9 to 16.7] | 3.6 [0.3 to 6.9]
  Maximum Change | 57.5 [50.9 to 64.1] | 33.1 [27.0 to 39.2]
Statistical Analysis 1: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Mean Change in ABPM heart rate; Mean Difference (Final Values) = 9.7, 95% CI 2-sided [7.4 to 12.0]
Statistical Analysis 2: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Maximum Change in ABPM heart rate; Mean Difference (Final Values) = 24.4, 95% CI 2-sided [17.9 to 30.9]

2. Secondary Outcome: Maximum and Mean Change From Baseline in Ambulatory Systolic and Diastolic Blood Pressure During Treatment With 18-mg LY2216684 or Placebo on Day 1
Description: Blood pressure (BP) was determined with ABPM. Mean pre-dose ABPM values from Day 1 in Period 1 were used as baseline. Changes in ABPM BP were determined from a 24-hour continuous ABPM monitoring for Day 1. LS mean changes from baseline were calculated with a mixed effects model including sequence, period, study day, treatment groups, and interaction between treatment groups and study day as fixed effects, and subject as random effect.
Time Frame: Baseline through the 24-hour interval on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeter of mercury (mm Hg)
Units Other Than Participants: Observations
Arm/Group | 18-mg LY2216684 | Placebo
Number analyzed (Participants) | 23 | 23
Number analyzed (Observations) | 23 | 27
millimeter of mercury (mm Hg)
  Mean Change, Systolic BP | 3.0 [-0.2 to 6.1] | -3.4 [-6.3 to -0.4]
  Maximum Change, Systolic BP | 28.8 [24.6 to 33.1] | 21.8 [17.9 to 25.6]
  Mean Change, Diastolic BP | 0.8 [-1.6 to 3.2] | -4.7 [-7.0 to -2.4]
  Maximum Change, Diastolic BP | 24.3 [21.0 to 27.7] | 18.7 [15.6 to 21.7]
Statistical Analysis 1: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Mean Change in ABPM systolic BP; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [3.9 to 8.8]
Statistical Analysis 2: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis — P-value is for the Maximum Change in ABPM systolic BP; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [2.6 to 11.6]
Statistical Analysis 3: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Mean Change in ABPM diastolic BP; Mean Difference (Final Values) = 5.51, 95% CI 2-sided [3.81 to 7.21]
Statistical Analysis 4: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — P-value is for the Maximum Change in ABPM diastolic BP; Mean Difference (Final Values) = 5.66, 95% CI 2-sided [2.13 to 9.20]

3. Secondary Outcome: Maximum and Mean Change From Baseline in Ambulatory Systolic and Diastolic Blood Pressure During Treatment With 18-mg LY2216684 or Placebo on Day 4
Description: BP was determined with ABPM. Mean pre-dose ABPM values from Day 1 in Period 1 were used as baseline. Changes in ABPM BP were determined from a 24-hour continuous ABPM monitoring for Day 4. LS mean changes from baseline were calculated with a mixed effects model including sequence, period, study day, treatment groups, and interaction between treatment groups and study day as fixed effects, and subject as random effect.
Time Frame: Baseline through the 24-hour interval on Day 4
Population: All participants with a baseline observation and at least 1 post-baseline observation on Day 4 were included in the analyses. Observations with 18-mg LY2216684 included Periods 1 and 2. Observations with Placebo included Periods 1, 2, and 3. Therefore, some participants contributed 2 Placebo observations to the overall data.
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeter of mercury (mm Hg)
Units Other Than Participants: Observations
Arm/Group | 18-mg LY2216684 | Placebo
Number analyzed (Participants) | 22 | 23
Number analyzed (Observations) | 22 | 27
millimeter of mercury (mm Hg)
  Mean Change, Systolic BP | -0.3 [-3.4 to 2.8] | -3.2 [-6.2 to -0.2]
  Maximum Change, Systolic BP | 24.1 [19.9 to 28.4] | 21.4 [17.6 to 25.3]
  Mean Change, Diastolic BP | 0.04 [-2.4 to 2.4] | -5.1 [-7.4 to -2.8]
  Maximum Change, Diastolic BP | 22.6 [19.3 to 26.0] | 16.1 [13.0 to 19.2]
Statistical Analysis 1: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0224, Mixed Models Analysis — P-value is for the Mean Change in ABPM systolic BP; Mean Difference (Final Values) = 2.90, 95% CI 2-sided [0.418 to 5.38]
Statistical Analysis 2: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.2453, Mixed Models Analysis — P-value is for the Maximum Change in ABPM systolic BP; Mean Difference (Final Values) = 2.70, 95% CI 2-sided [-1.88 to 7.29]
Statistical Analysis 3: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value if for the Mean Change in ABPM diastolic BP; Mean Difference (Final Values) = 5.10, 95% CI 2-sided [3.37 to 6.82]
Statistical Analysis 4: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — P-value is for the Maximum Change in ABPM diastolic BP; Mean Difference (Final Values) = 6.53, 95% CI 2-sided [2.95 to 10.1]

4. Secondary Outcome: Maximum and Mean Change From Baseline in ABPM Heart Rate During Treatment With 36-mg LY2216684 or Placebo on Day 4
Description: Heart rate was determined with ABPM. Mean pre-dose ABPM values from Day 1 in Period 1 were used as baseline. Changes in ABPM heart rate were determined from a 24-hour continuous ABPM monitoring for Day 4. LS mean changes from baseline were calculated with a mixed effects model including sequence, period, study day, treatment groups, and interaction between treatment groups and study day as fixed effects, and subject as random effect.
Time Frame: Baseline through the 24-hour interval on Day 4
Population: All participants with a baseline observation and at least 1 post-baseline observation on Day 4 were included in the analyses. Observations with 36-mg LY2216684 included Period 3. Observations with Placebo included Periods 1, 2, and 3. Therefore, some participants contributed 2 Placebo observations to the overall data.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Units Other Than Participants: Observations
Groups:
- 36-mg LY2216684: Participants received a single, oral dose of 36-mg LY2216684 each day over 4 days.
Arm/Group | 36-mg LY2216684 | Placebo
Number analyzed (Participants) | 18 | 23
Number analyzed (Observations) | 18 | 27
beats per minute (bpm)
  Mean Change | 15.8 [11.8 to 19.7] | 3.0 [-0.3 to 6.3]
  Maximum Change | 54.1 [45.4 to 62.7] | 31.1 [25.0 to 37.2]
Statistical Analysis 1: Comparison: 36-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Mean Change in ABPM heart rate; Mean Difference (Final Values) = 12.8, 95% CI 2-sided [8.7 to 16.9]
Statistical Analysis 2: Comparison: 36-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — P-value is for the Maximum Change in ABPM heart rate; Mean Difference (Final Values) = 23.0, 95% CI 2-sided [11.4 to 34.5]

5. Secondary Outcome: Maximum and Mean Change From Baseline in ABPM Systolic and Diastolic Blood Pressure During Treatment With 36-mg LY2216684 or Placebo on Day 4
Description: as for outcome 3
Time Frame: Baseline through the 24-hour interval on Day 4
Population: as for outcome 4
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeter of mercury (mm Hg)
Units Other Than Participants: Observations
Arm/Group | 36-mg LY2216684 | Placebo
Number analyzed (Participants) | 18 | 23
Number analyzed (Observations) | 18 | 27
millimeter of mercury (mm Hg)
  Mean Change, Systolic BP | -0.4 [-4.2 to 3.4] | -3.2 [-6.2 to -0.2]
  Maximum Change, Systolic BP | 29.0 [23.2 to 34.7] | 21.4 [17.6 to 25.3]
  Mean Change, Diastolic BP | -1.5 [-4.3 to 1.4] | -5.1 [-7.4 to -2.8]
  Maximum Change, Diastolic BP | 16.6 [12.1 to 21.2] | 16.1 [13.0 to 19.2]
Statistical Analysis 1: Comparison: 36-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.2120, Mixed Models Analysis — P-value is for the Mean Change in ABPM Systolic BP; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-1.6 to 7.2]
Statistical Analysis 2: Comparison: 36-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0640, Mixed Models Analysis — P-value is for the Maximum Change in ABPM Systolic BP; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [-0.4 to 15.5]
Statistical Analysis 3: Comparison: 36-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.0211, Mixed Models Analysis — P-value is for the Mean Change in ABPM Diastolic BP; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [0.5 to 6.7]
Statistical Analysis 4: Comparison: 36-mg LY2216684 vs Placebo; Test type: Superiority or Other; p = 0.8719, Mixed Models Analysis — P-value is for the Maximum Change in ABPM Diastolic BP; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-5.7 to 6.8]

6. Secondary Outcome: Maximum and Mean Change From Baseline in ABPM Heart Rate During Treatment With 18-mg LY2216684 or 36-mg LY2216684 on Day 4
Description: as for outcome 4
Time Frame: Baseline through the 24-hour interval on Day 4
Population: All participants with a baseline observation and at least 1 post-baseline observation on Day 4 were included in the analyses.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | 18-mg LY2216684 | 36-mg LY2216684
Number analyzed (Participants) | 22 | 18
beats per minute (bpm)
  Mean Change | 16.6 [13.2 to 20.1] | 15.8 [11.8 to 19.7]
  Maximum Change | 58.7 [52.1 to 65.4] | 54.1 [45.4 to 62.7]
Statistical Analysis 1: Comparison: 18-mg LY2216684 vs 36-mg LY2216684; Test type: Superiority or Other; p = 0.7133, Mixed Models Analysis — P-value is for the Mean Change in ABPM heart rate; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.3 to 3.7]
Statistical Analysis 2: Comparison: 18-mg LY2216684 vs 36-mg LY2216684; Test type: Superiority or Other; p = 0.4638, Mixed Models Analysis — P-value is for the Maximum Change in ABPM heart rate; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-17.2 to 7.9]

7. Primary Outcome: Maximum and Mean Change From Baseline in Ambulatory Heart Rate on Day 4
Description: Heart rate was determined during ABPM. Mean pre-dose ABPM values from Day 1 in Period 1 were used as baseline. Maximum and mean changes in ABPM heart rate were determined from 24 hour continuous ABPM monitoring for Day 4 (0 to 24 hours). LS mean changes from baseline were calculated with a mixed effects model including sequence, period, study day, treatment groups, and interaction between treatment groups and study day as fixed effects, and subject as random effect.
Time Frame: Baseline through the 24-hour interval on Day 4
Population: All participants with a baseline observation and at least 1 post-baseline observation on Day 4 were included in the analyses. Observations with 18-mg LY2216684 were made in Periods 1 and 2. Observations with Placebo included Periods 1, 2, and 3. Therefore, some participants contributed 2 Placebo observations to the overall data.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Units Other Than Participants: Observations
Arm/Group | 18-mg LY2216684 | Placebo
Number analyzed (Participants) | 22 | 23
Number analyzed (Observations) | 22 | 27
beats per minute (bpm)
  Mean Change | 16.6 [13.2 to 20.1] | 3.0 [-0.3 to 6.3]
  Maximum Change | 58.7 [52.1 to 65.4] | 31.1 [25.0 to 37.2]
Statistical Analysis 1: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Mean Change in ABPM heart rate; Mean Difference (Final Values) = 13.6, 95% CI 2-sided [11.3 to 15.9]
Statistical Analysis 2: Comparison: 18-mg LY2216684 vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value is for the Maximum Change in ABPM heart rate; Mean Difference (Final Values) = 27.6, 95% CI 2-sided [21.1 to 34.2]

8. Secondary Outcome: Maximum and Mean Change From Baseline in ABPM Systolic and Diastolic Blood Pressure During Treatment With 18-mg LY2216684 or 36-mg LY2216684 on Day 4
Description: as for outcome 3
Time Frame: Baseline through the 24-hour interval on Day 4
Population: as for outcome 6
Measure: Least Squares Mean (90% Confidence Interval); unit: millimeter of mercury (mm Hg)
Arm/Group | 18-mg LY2216684 | 36-mg LY2216684
Number analyzed (Participants) | 22 | 18
millimeter of mercury (mm Hg)
  Mean Change, Systolic BP | -0.3 [-3.4 to 2.8] | -0.4 [-4.2 to 3.4]
  Maximum Change, Systolic BP | 24.1 [19.9 to 28.4] | 29.0 [23.2 to 34.7]
  Mean Change, Diastolic BP | 0.04 [-2.4 to 2.4] | -1.5 [-4.3 to 1.4]
  Maximum Change, Diastolic BP | 22.6 [19.3 to 26.0] | 16.6 [12.1 to 21.2]
Statistical Analysis 1: Comparison: 18-mg LY2216684 vs 36-mg LY2216684; Test type: Superiority or Other; p = 0.9609, Mixed Models Analysis — P-value is for the Mean Change in ABPM Systolic BP; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-4.9 to 4.7]
Statistical Analysis 2: Comparison: 18-mg LY2216684 vs 36-mg LY2216684; Test type: Superiority or Other; p = 0.2731, Mixed Models Analysis — P-value is for the Maximum Change in ABPM Systolic BP; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-3.9 to 13.6]
Statistical Analysis 3: Comparison: 18-mg LY2216684 vs 36-mg LY2216684; Test type: Superiority or Other; p = 0.3779, Mixed Models Analysis — P-value is for the Mean Change in ABPM Diastolic BP; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.8 to 1.8]
Statistical Analysis 4: Comparison: 18-mg LY2216684 vs 36-mg LY2216684; Test type: Superiority or Other; p = 0.0828, Mixed Models Analysis — P-value is for the Maximum Change in ABPM Diastolic BP; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-12.8 to 0.8]

ADVERSE EVENTS:
Time Frame: Periods 1, 2, and 3 through 7-day follow-up
Arm/Group | 18-mg LY2216684 | 36-mg LY2216684 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/19 | 0/24
Other Adverse Events (participants affected / at risk) | 20/24 | 12/19 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18-mg LY2216684 (N=24) | 36-mg LY2216684 (N=19) | Placebo (N=24)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 18-mg LY2216684 (N=24) | 36-mg LY2216684 (N=19) | Placebo (N=24)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 9 (9) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (4)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (4)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1/15 (1) | 0/12 (0) | 0/15 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0/15 (0) | 0/12 (0) | 1/15 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days